CLINICAL TRIAL: NCT04172701
Title: CITRUS Study (Comparing the Incidence Between Tiotropium and ICS/LABA in Real World Use in South Korea)
Brief Title: A Study in South Korea Using Medical Records to Look at Different Treatments for Chronic Obstructive Airway Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0205-0542
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LAMA: Chronic obstructive pulmonary disease (COPD) patients who were prescribed long-acting muscarinic antagonists (LAMA) monotherapy between 01 January 2005 and 30 April 2015.
  Interventions: Drug: Long-acting Muscarinic Antagonists (LAMA)
- ICS/LABA: Chronic obstructive pulmonary disease (COPD) patients who were prescribed a fixed-dose combination (FDC) of inhaled corticosteroid (ICS)/long-acting beta agonists (LABA) between 01 January 2005 and 30 April 2015.
  Interventions: Drug: Inhaled corticosteroid (ICS)/Long-acting Beta Agonists (LABA)

INTERVENTIONS:
Drug: Long-acting Muscarinic Antagonists (LAMA) — drug
  Groups: LAMA
Drug: Inhaled corticosteroid (ICS)/Long-acting Beta Agonists (LABA) — drug
  Groups: ICS/LABA

SUMMARY:
Non-interventional, Single-country study based on existing data from medical records of COPD patients treated with LAMA or fixed dose combination of ICS/LABA

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD [based on ICD-10 code(J43.x-44.x except J430), as the primary or within the fourth secondary diagnosis and initiated LAMA or ICS/LABA more than twice a year from Jan 1, 2005 to Apr 30 2016].
* Age >55 years old

Exclusion Criteria:

* Prescription history with any long acting bronchodilator for maintenance therapy (the patient should be inhaler naïve)
* Prescription history with ipratropium bromide
* Prescription history with Leukotriene receptor antagonist(LTRA) or ICS
* Patients with lung cancer, IPF, ILD or lung transplantation at the time of COPD diagnosis

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic obstrutive pulmonary disease
Sampling Method: Probability Sample
Enrollment: 9284 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a retrospective, observational, non-interventional cohort study using national health insurance claims data from the National Health Insurance Service (NHIS) of South Korea to compare the real-world outcomes among chronic obstructive pulmonary disease (COPD) patients initiating long-acting muscarinic antagonists (LAMA) or inhaled corticosteroid (ICS)/long-acting beta agonists (LABA) in South Korea.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included.
Period: Overall Study
Arm/Group | LAMA | ICS/LABA
Started | 6352 | 2932
Propensity Score (PS) Matched Population | 2444 | 2444
Completed | 6352 | 2932
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score matching population: To address the imbalance of potential confounders between LAMA and ICS/LABA groups, treatment groups were matched using propensity scores estimated as by multiple logistic regression analysis based on age, sex, socioeconomics status, Charlson Comorbidity Index, asthma and history of chronic obstructive pulmonary disease (COPD) exacerbation.
Groups:
- Total: Total of all reporting groups
Arm/Group | LAMA | ICS/LABA | Total
Number analyzed (Participants) | 2444 | 2444 | 4888
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.57 (7.85) | 69.73 (7.91) | 69.65 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 590 | 622 | 1212
  Male | 1854 | 1822 | 3676
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate for the First Pneumonia Event
Description: Pneumonia was defined as ≥1 inpatient or outpatient claims 1) with ICD-10 codes for pneumonia recorded as any diagnosis in inpatient claims or primary ~ 4th secondary diagnosis in outpatient claims, AND 2) with diagnostic test code for chest-X ray or chest- computed tomography (CT), AND 3) with antibiotics prescription during the following period after the index date. To assess the incidence of pneumonia event, the first pneumonia event observed during the follow-up period was considered.
  Incidence rate for the first pneumonia event was calculated as below:
  Incidence rate per 1000 person-years= Number of patients with event/ sum of event-free period during the follow-up period (1000 person-years)
Time Frame: From the index date (i.e. between 01 January 2005 and 30 April 2015) up to the earliest of discontinuation of the index drug (i.e. LAMA or ICS/LABA), death, or 30 April 2016 (i.e. cut-off date for data retrieving), up to 136 months.
Population: as for baseline characteristics
Measure: Number; unit: patients/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
patients/1000 person-years | 109.82 | 167.10
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual log-linked Poisson model

2. Primary Outcome: Incidence Rate of Pneumonia Events
Description: Pneumonia was defined as ≥1 inpatient or outpatient claims 1) with ICD-10 codes for pneumonia recorded as any diagnosis in inpatient claims or primary ~ 4th secondary diagnosis in outpatient claims, AND 2) with diagnostic test code for chest-X ray or chest- computed tomography (CT), AND 3) with antibiotics prescription during the following period after the index date.
  This outcome measure reports: Total number of pneumonia events/ sum of follow-up duration (person-years) for all participants
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: events/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
events/1000 person-years | 182.51 | 264.99
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.001, Individual t-test or Wilcoxon test

3. Primary Outcome: Time to First Pneumonia Event From the Index Date
Description: Pneumonia was defined as ≥1 inpatient or outpatient claims 1) with ICD-10 codes for pneumonia recorded as any diagnosis in inpatient claims or primary ~ 4th secondary diagnosis in outpatient claims, AND 2) with diagnostic test code for chest-X ray or chest- computed tomography (CT), AND 3) with antibiotics prescription during the following period after the index date. Date of pneumonia event was defined as the starting date of outpatient claim, or as the admission date of inpatient claim with the above 3 conditions to define pneumonia event.
  Mean and Standard Deviation of time to first pneumonia event from the index date was estimated using the Kaplan-Meier curve.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
days | 544.96 (609.83) | 413.35 (475.8)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Log Rank

4. Primary Outcome: Number of Patients With Pneumonia Event
Description: Pneumonia was defined as ≥1 inpatient or outpatient claims 1) with ICD-10 codes for pneumonia recorded as any diagnosis in inpatient claims or primary ~ 4th secondary diagnosis in outpatient claims, AND 2) with diagnostic test code for chest-X ray or chest- computed tomography (CT), AND 3) with antibiotics prescription during the following period after the index date.
  Number of patients with pneumonia event is reported.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
Participants | 501 | 605
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; The Cox proportional hazards regression took into account the fact that individual matching (1:1) was performed by considering the exposed patient and his/her matched control as one stratum and including this as a stratum in the Cox proportional hazards model.The presented Hazard Ratio (HR) was estimated using the LAMA as a reference group; Test type: Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 1.475, 95% CI 2-sided [1.308 to 1.663]

5. Primary Outcome: Incidence Rate of the First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Event (All Types)
Description: To assess the incidence of COPD exacerbation event (all types), the first COPD exacerbation event among pre-defined moderate COPD exacerbation and severe COPD exacerbation event observed within the 12-month period after the index date was considered.
  Moderate COPD exacerbation was defined as ≥ 1 outpatient claims 1) with ICD-10 codes for COPD recorded as primary ~ 4th secondary diagnosis, AND 2) with systemic steroids and/or antibiotics prescription within 12 months after the index date. Severe COPD exacerbation was defined as ≥ 1 Emergency Room (ER) visit or inpatient claims 1) with ICD-10 codes for COPD or diseases due to COPD worsening as any diagnosis, AND 2) with systemic steroids and/or antibiotics prescription.
  Incidence rate of COPD exacerbation events (all types) was calculated as below: Incidence rate per 1000 person-years= Number of patients with event/sum of event-free period during the follow-up period (1000 person-years)
Time Frame: Up to 12 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Number; unit: patients/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
patients/1000 person-years | 714.18 | 827.77
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0003, Individual log-linked Poisson model

6. Primary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Events (All Types)
Description: To assess the frequency of all types (moderate and severe) COPD exacerbation events, any events observed within the 12-month period after the index date was considered.
  Moderate COPD exacerbation was defined as ≥ 1 outpatient claims 1) with ICD-10 codes for COPD recorded as primary ~ 4th secondary diagnosis, AND 2) with systemic steroids and/or antibiotics prescription within 12 months after the index date. Severe COPD exacerbation was defined as ≥ 1 Emergency Room (ER) visit or inpatient claims 1) with ICD-10 codes for COPD or diseases due to COPD worsening as any diagnosis, AND 2) with systemic steroids and/or antibiotics prescription.
  Outcome measure reports: Total number of COPD exacerbation events (all types)/sum of follow-up duration (person-years) for all participants
Time Frame: Up to 12 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Number; unit: events/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
events/1000 person-years | 1357.48 | 1523.68
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.001, Individual t-test or Wilcoxon test

7. Primary Outcome: Number of Patients With Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Events
Description: Number of patients with Chronic Obstructive Pulmonary Disease (COPD) exacerbation (moderate or severe) events is reported.
  Moderate COPD exacerbation was defined as ≥ 1 outpatient claims 1) with ICD-10 codes for COPD recorded as primary ~ 4th secondary diagnosis, AND 2) with systemic steroids and/or antibiotics prescription within 12 months after the index date. Severe COPD exacerbation was defined as ≥ 1 Emergency Room (ER) visit or inpatient claims 1) with ICD-10 codes for COPD or diseases due to COPD worsening as any diagnosis, AND 2) with systemic steroids and/or antibiotics prescription.
Time Frame: Up to 12 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
Participants | 1170 | 1285
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; The Cox proportional hazards regression took into account the fact that individual matching (1:1) was performed by considering the exposed patient and his/her matched control as one stratum and including this as a stratum in the Cox proportional hazards model. The presented Hazard Ratio (HR) was estimated using the LAMA as a reference group; Test type: Other; p = 0.0006, Regression, Cox; Hazard Ratio (HR) = 1.145, 95% CI 2-sided [1.059 to 1.237]

8. Primary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Event From the Index Date
Description: Mean and Standard Deviation of time to first COPD exacerbation (moderate or severe) event from the index date was estimated using the Kaplan-Meier curve.
  Moderate COPD exacerbation was defined as ≥ 1 outpatient claims 1) with ICD-10 codes for COPD recorded as primary ~ 4th secondary diagnosis, AND 2) with systemic steroids and/or antibiotics prescription within 12 months after the index date. Severe COPD exacerbation was defined as ≥ 1 Emergency Room (ER) visit or inpatient claims 1) with ICD-10 codes for COPD or diseases due to COPD worsening as any diagnosis, AND 2) with systemic steroids and/or antibiotics prescription. Date of severe COPD exacerbation event was defined as the starting date of ER claims or admission date of inpatient claims with the above 2 conditions to define moderate COPD exacerbation event.
Time Frame: Up to 12 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
days | 113.94 (106.08) | 111.92 (105.04)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.00074, Log Rank

9. Primary Outcome: Incidence Rate of Initiating Triple Combination Therapy
Description: To assess the incidence rate of initiating triple combination therapy, the first triple combination therapy observed during the follow-up period was considered.
  Triple combination therapy of inhaled corticosteroids (ICS), long-acting beta agonists (LABA) and long-acting muscarinic antagonists (LAMA) was defined as ≥ 1 outpatient or inpatient claims with a combination of ICS, LABA, and LAMA. Three components of ICS, LABA and LAMA MUST have been prescribed together in a same prescription issued on same date to be considered as triple combination therapy (i.e. ICS/LABA fixed dose combination (FDC) and LAMA, ICS and LABA/LAMA FDC, ICS/LABA FDC and LABA/LAMA FDC, ICS and LABA and LAMA are all considered as triple combination therapy).
  Incidence rate of initiating triple combination therapy is reported as: Incidence rate per 1000 person-years= Number of patients with event/ sum of event-free period during the follow-up period (1000 person-years)
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: patients/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
patients/1000 person-years | 80.98 | 139.82
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual log-linked Poisson model

10. Primary Outcome: Number of Patients Who Initiated a Triple Combination Therapy
Description: Number of patients who initiated a triple combination therapy is reported. Triple combination therapy of inhaled corticosteroids (ICS), long-acting beta agonists (LABA) and long-acting muscarinic antagonists (LAMA) was defined as ≥ 1 outpatient or inpatient claims with a combination of ICS, LABA, and LAMA. Three components of ICS, LABA and LAMA MUST have been prescribed together in a same prescription issued on same date to be considered as triple combination therapy (i.e. ICS/LABA fixed dose combination (FDC) and LAMA, ICS and LABA/LAMA FDC, ICS/LABA FDC and LABA/LAMA FDC, ICS and LABA and LAMA are all considered as triple combination therapy).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
Participants | 383 | 518
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 1.601, 95% CI 2-sided [1.404 to 1.826]

11. Primary Outcome: Time to Initiating Triple Combination Therapy From the Index Date
Description: Median and Inter-Quartile Range of time to initiating triple combination therapy from the index date was estimated using the Kaplan-Meier curve.
  Triple combination therapy of inhaled corticosteroids (ICS), long-acting beta agonists (LABA) and long-acting muscarinic antagonists (LAMA) was defined as ≥ 1 outpatient or inpatient claims with a combination of ICS, LABA, and LAMA. Three components of ICS, LABA and LAMA MUST have been prescribed together in a same prescription issued on same date to be considered as triple combination therapy (i.e. ICS/LABA fixed dose combination (FDC) and LAMA, ICS and LABA/LAMA FDC, ICS/LABA FDC and LABA/LAMA FDC, ICS and LABA and LAMA are all considered as triple combination therapy).
  Date of triple combination therapy was defined as the starting date of outpatient claim or admission date of inpatient claim with a combination of ICS/LABA and LAMA.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
days | 281 [92 to 606] | 207 [99 to 394]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Log Rank

12. Secondary Outcome: All-cause Healthcare Resource Utilization (HCRU): Number of Any Medical Visit (Per Person Per Month)
Description: Mean and Standard Deviation of any medical visit per person per month is reported. Medical visits were calculated as the sum of inpatient and outpatient visits assuming that emergency room (ER) visits, intensive care unit (ICU) visits and visit for pharmacy dispensation would be counted with the inclusion of inpatient and outpatient visit.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 2.81 (2.30) | 2.73 (1.93)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.2875, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: All-cause Healthcare Resource Utilization (HCRU): Number of Outpatient Visits (Per Person Per Month)
Description: Mean and Standard Deviation of outpatient visits per person per month is reported. Outpatient visit was defined as clinic, hospital, or other medical institution (e.g. public health, etc.) visit as an outpatient.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 2.75 (2.29) | 2.66 (1.92)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.4602, Individual t-test or Wilcoxon test

14. Secondary Outcome: All-cause Healthcare Resource Utilization (HCRU): Number of Inpatient Visits (Per Person Per Month)
Description: Mean and Standard Deviation of inpatient visits per person per month is reported. Inpatient visit was defined as at least 1 overnight stay in a hospital as an inpatient.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 0.06 (0.10) | 0.07 (0.13)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0062, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: All-cause Healthcare Resource Utilization (HCRU): Number of Emergency Room (ER) Visits (Per Person Per Month)
Description: Mean and Standard Deviation of ER visits per person per month is reported.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 0.03 (0.08) | 0.04 (0.09)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0002, Individual t-test or Wilcoxon test

16. Secondary Outcome: All-cause Healthcare Resource Utilization (HCRU): Number of Intensive Care Unit (ICU) Visits (Per Person Per Month)
Description: Mean and Standard Deviation of ICU visits per person per month is reported.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 0.00 (0.02) | 0.01 (0.02)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.4907, Individual t-test or Wilcoxon test

17. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Resource Utilization (HCRU): Number of Any Medical Visit (Per Person Per Month)
Description: COPD-related HCRU was defined as medical claims with ICD-10 codes for COPD and/or COPD-related diseases. Mean and Standard Deviation of any medical visit (inpatient and outpatient visits which include emergency room (ER) and intensive care unit (ICU) visits) per person per month is reported. For outpatient claims, COPD-related HCRU was defined as claims with ICD-10 codes for COPD as primary ~ 4th secondary diagnosis. For inpatient claims, COPD-related HCRU was defined as claims with ICD-10 codes for COPD and/or for diseases due to COPD worsening as any diagnosis.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 0.66 (0.39) | 0.60 (0.47)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.001, Individual t-test or Wilcoxon test

18. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Resource Utilization (HCRU): Number of Outpatient Visits (Per Person Per Month)
Description: Mean and Standard Deviation of outpatient visits per person per month is reported. For outpatient claims, COPD-related HCRU was defined as claims with ICD-10 codes for COPD as primary ~ 4th secondary diagnosis.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 0.63 (0.38) | 0.56 (0.46)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Resource Utilization (HCRU): Number of Inpatient Visits (Per Person Per Month)
Description: Mean and Standard Deviation of inpatient visits per person per month is reported. For inpatient claims, COPD-related HCRU was defined as claims with ICD-10 codes for COPD and/or for diseases due to COPD worsening as any diagnosis.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 0.03 (0.07) | 0.03 (0.10)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.543, Individual t-test or Wilcoxon test

20. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Resource Utilization (HCRU): Number of Emergency Room (ER) (Visits Per Person Per Month)
Description: Mean and Standard Deviation of ER visits per person per month is reported.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 0.01 (0.03) | 0.01 (0.05)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.080, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Resource Utilization (HCRU): Number of Intensive Care Unit (ICU) Visits (Per Person Per Month)
Description: Mean and Standard Deviation of ICU visits per person per month is reported.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: visits per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
visits per person per month | 0.00 (0.01) | 0.00 (0.02)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.363, Individual t-test or Wilcoxon test

22. Secondary Outcome: All-cause Healthcare Costs: Total Medical Costs (Per Person Per Month)
Description: Mean and Standard Deviation of total medical costs per person per month is reported. Total medical costs were estimated as the sum of medical costs (inpatient + outpatient) and pharmacy dispensation costs (drug cost + pharmacy service cost). Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 441.08 (527.43) | 510.42 (619.59)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual t-test or Wilcoxon test

23. Secondary Outcome: All-cause Healthcare Costs: Hospitalization Costs (Per Person Per Month)
Description: Mean and Standard Deviation of hospitalization costs per person per month is reported. Hospitalization costs were estimated as the total costs of services from all inpatient claims (e.g. cost for procedure, diagnostic test, medication, patient meal, and bed stay, etc.). Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 176.26 (467.48) | 208.40 (558.44)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0494, Individual t-test or Wilcoxon test

24. Secondary Outcome: All-cause Healthcare Costs: Outpatient Medical Costs (Per Person Per Month)
Description: Mean and Standard Deviation of outpatient medical costs per person per month is reported. Outpatient medical costs were estimated as the total costs of services from all outpatient claims (e.g. cost for procedure, diagnostic test, prescription, physician fee, etc.). Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 92.44 (132.65) | 100.20 (147.37)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0091, Individual t-test or Wilcoxon test

25. Secondary Outcome: All-cause Healthcare Costs: Outpatient Pharmacy Dispensation Costs (Per Person Per Month)
Description: Mean and Standard Deviation of outpatient pharmacy dispensation costs per person per month is reported. Outpatient pharmacy dispensation costs were estimated as the total costs of services from all outpatient pharmacy claims (pharmacy dispensing service costs + medication costs). Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 172.38 (126.23) | 201.81 (156.85)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual t-test or Wilcoxon test

26. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Costs: Total Medical Costs (Per Person Per Month)
Description: Mean and Standard Deviation of COPD-related total medical costs per person per month is reported. COPD-related total medical costs were estimated as the sum of medical costs (inpatient + outpatient) of medical claims with ICD-10 codes for COPD and/or COPD-related diseases and pharmacy dispensation costs (drug costs + pharmacy service costs) of pharmacy claims including dispensation of ICS/LABA, LABA, LAMA, LABA/LAMA, short-acting beta-2 agonist (SABAs), short-acting muscarinic antagonist (SAMAs), SABA/SAMA, theophlliyne, or Phosphodiesterase-4 (PDE4) inhibitor. Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 243.82 (408.63) | 295.83 (528.06)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual t-test or Wilcoxon test

27. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Costs: Hospitalization Costs (Per Person Per Month)
Description: Mean and Standard Deviation of COPD-related hospitalization costs per person per month is reported. COPD-related hospitalization costs were estimated as the total costs of services (e.g. costs for procedure, diagnostic test, medication, patient meal, and bed stay, etc.) from all inpatient claims (medical claims with ICD-10 codes for COPD and/or for diseases due to COPD worsening as any diagnosis).
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 112.87 (380.37) | 132.22 (491.24)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.7298, Individual t-test or Wilcoxon test

28. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Costs: Outpatient Medical Costs (Per Person Per Month)
Description: Mean and Standard Deviation of COPD-related outpatient medical costs per person per month is reported. COPD-related outpatient medical costs were estimated as the total costs of services (e.g. costs for procedure, diagnostic test, prescription, physician fee, etc.) from all outpatient claims (medical claims with ICD-10 codes for COPD as primary ~ 4th secondary diagnosis).
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 21.19 (27.34) | 22.23 (36.53)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0093, Individual t-test or Wilcoxon test

29. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Costs: Outpatient Pharmacy Dispensation Costs (Per Person Per Month)
Description: Mean and Standard Deviation of COPD-related outpatient pharmacy dispensation costs per person per month is reported.
  COPD related outpatient pharmacy dispensation costs were estimated as the total costs of services (pharmacy dispensing service costs + medication costs) from all outpatient pharmacy claims (pharmacy claims including dispensation of ICS/LABA, LABA, LAMA, LABA/LAMA, short-acting beta-2 agonist (SABAs), short-acting muscarinic antagonist (SAMAs), SABA/SAMA, theophlliyne, or Phosphodiesterase-4 (PDE4) inhibitor).
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 109.75 (101.63) | 141.39 (137.40)
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual t-test or Wilcoxon test

30. Secondary Outcome: Adjusted All-cause Costs: Total Medical Costs (Per Person Per Month)
Description: Mean and 95% Confidence Interval of adjusted all-cause total medical costs per person per month is reported. All-cause total medical costs were adjusted for baseline characteristics and healthcare resource utilization (HCRU) and healthcare costs occurred during baseline period. Total medical cost were estimated as the sum of medical costs (inpatient + outpatient) and pharmacy dispensation costs (drug costs + pharmacy service costs).
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 403.08 [353.66 to 459.40] | 474.50 [415.29 to 542.16]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual t-test or Wilcoxon test; Cost ratio = 1.177, 95% CI 2-sided [1.104 to 1.255] — cost ratio = cost of ICS/LABA divided by cost of LAMA

31. Secondary Outcome: Adjusted All-cause Costs: Hospitalization Costs (Per Person Per Month)
Description: Mean and 95% Confidence Interval of adjusted all-cause hospitalization costs per person per month.
  All-cause hospitalization costs were estimated as the total costs of services from all inpatient claims (e.g. costs for procedure, diagnostic test, medication, patient meal, and bed stay, etc.) and were adjusted for baseline characteristics and healthcare resource utilization (HCRU) and healthcare costs occurred during baseline period.
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 236.65 [177.23 to 316.00] | 282.58 [209.20 to 381.70]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0103, Individual t-test or Wilcoxon test; Cost ratio = 1.194, 95% CI 2-sided [1.043 to 1.367] — cost ratio = cost of ICS/LABA divided by cost of LAMA

32. Secondary Outcome: Adjusted All-cause Costs: Outpatient Medical Costs (Per Person Per Month)
Description: Mean and 95% Confidence Interval of adjusted all-cause outpatient medical costs per person per month. All-cause outpatient medical costs were estimated as the total costs of services from all outpatient claims (e.g. costs for procedure, diagnostic test, prescription, physician fee, etc.) and were adjusted for baseline characteristics and healthcare resource utilization (HCRU) and healthcare costs occurred during baseline period.
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 77.41 [64.68 to 92.64] | 85.45 [71.88 to 101.58]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0030, Individual t-test or Wilcoxon test; Cost ratio = 1.104, 95% CI 2-sided [1.034 to 1.178] — cost ratio = cost of ICS/LABA divided by cost of LAMA

33. Secondary Outcome: Adjusted All-cause Costs: Outpatient Pharmacy Dispensation Costs (Per Person Per Month)
Description: Mean and 95% Confidence Interval of adjusted all-cause outpatient pharmacy dispensation costs per person per month is reported. All-cause outpatient pharmacy dispensation cost were estimated as the total costs of services from all outpatient pharmacy claims (pharmacy dispensing service costs + medication costs) and were adjusted for baseline characteristics and healthcare resource utilization (HCRU) and healthcare costs occurred during baseline period.
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 161.18 [148.87 to 174.52] | 189.32 [175.23 to 204.54]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual t-test or Wilcoxon test; Cost ratio = 1.175, 95% CI 2-sided [1.130 to 1.221] — cost ratio = cost of ICS/LABA divided by cost of LAMA

34. Secondary Outcome: Adjusted Chronic Obstructive Pulmonary Disease (COPD)-Related Costs: Total Medical Costs (Per Person Per Month)
Description: Mean and 95% Confidence Interval of adjusted COPD-related total medical costs per person per month is reported. COPD-related total medical costs were estimated as the sum of medical costs (inpatient + outpatient) of medical claims with ICD-10 codes for COPD and/or COPD-related diseases and pharmacy dispensation costs (drug costs + pharmacy service costs) of pharmacy claims including dispensation of ICS/LABA, LABA, LAMA, LABA/LAMA, short-acting beta-2 agonist (SABAs), short-acting muscarinic antagonist (SAMAs), SABA/SAMA, theophlliyne, or Phosphodiesterase-4 (PDE4) inhibitor and were adjusted for baseline characteristics and healthcare resource utilization (HCRU) and healthcare costs occurred during baseline period.
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 216.37 [189.65 to 246.85] | 267.32 [235.25 to 303.78]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual t-test or Wilcoxon test; Cost ratio = 1.236, 95% CI 2-sided [1.134 to 1.346] — cost ratio = cost of ICS/LABA divided by cost of LAMA

35. Secondary Outcome: Adjusted Chronic Obstructive Pulmonary Disease (COPD)-Related Costs: Hospitalization Costs (Per Person Per Month)
Description: Mean and 95% Confidence Interval of COPD-related hospitalization costs per person per month is reported.
  COPD-related hospitalization costs were estimated as the total costs of services (e.g. costs for procedure, diagnostic test, medication, patient meal, and bed stay, etc.) from all inpatient claims (medical claims with ICD-10 codes for COPD and/or for diseases due to COPD worsening as any diagnosis and were adjusted for baseline characteristics and healthcare resource utilization (HCRU) and healthcare costs occurred during baseline period.
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 178.25 [133.93 to 237.23] | 216.31 [162.45 to 288.01]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.0212, Individual t-test or Wilcoxon test; Cost ratio = 1.214, 95% CI 2-sided [1.029 to 1.431] — cost ratio = cost of ICS/LABA divided by cost of LAMA

36. Secondary Outcome: Adjusted Chronic Obstructive Pulmonary Disease (COPD)-Related Costs: Outpatient Medical Costs (Per Person Per Month)
Description: Mean and 95% Confidence Interval of COPD-related outpatient medical costs (per person per month) is reported. COPD-related outpatient medical costs were estimated as the total costs of services (e.g. costs for procedure, diagnostic test, prescription, physician fee, etc.) from all outpatient claims (medical claims with ICD-10 codes for COPD as primary ~ 4th secondary diagnosis) and were adjusted for baseline characteristics and healthcare resource utilization (HCRU) and healthcare costs occurred during baseline period.
  Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 20.20 [16.66 to 24.49] | 20.72 [16.91 to 25.38]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.5024, Individual t-test or Wilcoxon test; Cost ratio = 1.026, 95% CI 2-sided [0.952 to 1.105] — cost ratio = cost of ICS/LABA divided by cost of LAMA

37. Secondary Outcome: Adjusted Chronic Obstructive Pulmonary Disease (COPD)-Related Costs: Outpatient Pharmacy Dispensation Costs (Per Person Per Month)
Description: Mean and 95% Confidence Interval of COPD-related outpatient pharmacy dispensation costs (per person per month) is reported. COPD related outpatient pharmacy dispensation costs were estimated as the total costs of services (pharmacy dispensing service costs + medication costs) from all outpatient pharmacy claims (pharmacy claims including dispensation of ICS/LABA, LABA, LAMA, LABA/LAMA, short-acting beta-2 agonist (SABAs), short-acting muscarinic antagonist (SAMAs), SABA/SAMA, theophlliyne, or Phosphodiesterase-4 (PDE4) inhibitor) and were adjusted for baseline characteristics and healthcare resource utilization (HCRU) and healthcare costs occurred during baseline period Costs were converted to US dollars using the average 2019 exchange rate: US$ = 1166.51 KRW (South Korean won) and were also adjusted to calendar year 2019 using the Consumer Price Index of South Korea.
Time Frame: Up to 36 months from the index date. Index date was between 01 January 2005 and 30 April 2015.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars per person per month
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
dollars per person per month | 112.35 [102.68 to 122.92] | 146.53 [134.35 to 159.82]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p < 0.0001, Individual t-test or Wilcoxon test; Cost ratio = 1.304, 95% CI 2-sided [1.243 to 1.369] — cost ratio = cost of ICS/LABA divided by cost of LAMA

38. Secondary Outcome: Incidence Rate of All-cause Death
Description: Date of death event was defined as the date of death recorded in the National Health Information Database (NHID).
  Incidence rate of all-cause death was calculated as below: Incidence rate per 1000 person-years= Number of patients with event/ sum of event-free period during the follow-up period (1000 person-years)
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: patients/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
patients/1000 person-years | 9.38 | 10.09
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.7198, Individual log-linked Poisson model

39. Secondary Outcome: Number of Patients With the Event All-cause Death
Description: Number of patients with the event all-cause death is reported.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
Participants | 51 | 46
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.7341, Regression, Cox; Hazard Ratio (HR) = 1.072, 95% CI 2-sided [0.719 to 1.598]

40. Secondary Outcome: Time to Death From the Index Date
Description: Median and Inter-Quartile Range of time to death from the index date is reported. Date of death event was defined as the date of death recorded in the National Health Information Database (NHID). Time to death was estimated from the Kaplan-Meier curve.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
days | 609 [308 to 1070] | 350 [303 to 965]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.74, Log Rank

41. Secondary Outcome: Incidence Rate of Tuberculosis (TB) Event
Description: Tuberculosis (TB) was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for pulmonary TB recorded as any diagnosis, AND 2) with special benefit costs for TB patients during the following period after the index date. To assess the incidence of TB event, the first TB event observed during the follow-up period was considered. Incidence rate of TB was calculated as below:
  Incidence rate per 1000 person-years= Number of patients with event/ sum of event-free period during the follow-up period (1000 person-years)
Time Frame: From the index date (i.e. between 01 January 2005 and 30 April 2015) up to the earliest of discontinuation of the index drug (i.e. LAMA or ICS/LABA), death, or 30 April 2016 (i.e. study end date), up to 136 months.
Population: as for baseline characteristics
Measure: Number; unit: patients/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
patients/1000 person-years | 10.46 | 10.46
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.9985, Individual log-linked Poisson model

42. Secondary Outcome: Number of Patients With Tuberculosis (TB)
Description: Tuberculosis (TB) was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for pulmonary TB recorded as any diagnosis, AND 2) with special benefit costs for TB patients during the following period after the index date. Number of patients with tuberculosis (TB) is reported.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
Participants | 56 | 47
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.5097, Regression, Cox; Hazard Ratio (HR) = 0.879, 95% CI 2-sided [0.600 to 1.289]

43. Secondary Outcome: Time to First Tuberculosis (TB) Event From the Index Date
Description: Median and Inter-Quartile Range of time to first tuberculosis (TB) event is reported. Tuberculosis (TB) was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for pulmonary TB recorded as any diagnosis, AND 2) with special benefit costs for TB patients during the following period after the index date. Date of TB was defined as the admission date of inpatient claim or the starting date of outpatient claim with the above 2 conditions to define TB event. Median and Inter-Quartile Range of time to first tuberculosis (TB) event was estimated using the Kaplan-Meier curve.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
days | 1 [1 to 116.5] | 86 [1 to 318]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.51, Log Rank

44. Secondary Outcome: Incidence Rate of Lung Cancer
Description: Lung cancer was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for lung cancer recorded as any diagnosis, AND 2) with costs for patients with cancers during the following period after the index date. To assess the incidence of lung cancer event, the first lung cancer event observed during the follow-up period was considered.
  Incidence rate of lung cancer was calculated as below:
  Incidence rate per 1000 person-years= Number of patients with event/ sum of event-free period during the follow-up period (1000 person-years)
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: patients/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
patients/1000 person-years | 10.64 | 11.74
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.6069, Individual log-linked Poisson model

45. Secondary Outcome: Number of Patients With Lung Cancer
Description: Number of patients with lung cancer is reported. Lung cancer was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for lung cancer recorded as any diagnosis, AND 2) with costs for patients with cancers during the following period after the index date.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
Participants | 57 | 53
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.8960, Regression, Cox; Hazard Ratio (HR) = 1.025, 95% CI 2-sided [0.705 to 1.490]

46. Secondary Outcome: Time to Occurrence of Lung Cancer From the Index Date
Description: Median and Inter-Quartile Range of time to occurrence of lung cancer from the index date.
  Lung cancer was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for lung cancer recorded as any diagnosis, AND 2) with costs for patients with cancers during the following period after the index date.
  Date of lung cancer diagnosis was defined as the admission date of inpatient claim or the starting date of outpatient claim with the above 2 conditions to define lung cancer event.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
days | 91 [1 to 399] | 231 [77 to 600]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.9, Log Rank

47. Secondary Outcome: Incidence Rate of Non-tuberculosis Mycobacteria (NTM) Lung Disease
Description: Non-tuberculosis mycobacteria (NTM) lung disease was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for NTM recorded as any diagnosis during the following period after the index date. To assess the incidence of NTM event, the first NTM event observed during the follow-up period was considered.
  Incidence rate of NTM lung disease was calculated as below:
  Incidence rate per 1000 person-years= Number of patients with event/ sum of event-free period during the follow-up period (1000 person-years)
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: patients/1000 person-years
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
patients/1000 person-years | 5.00 | 3.09
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.1354, Individual log-linked Poisson model

48. Secondary Outcome: Number of Patients With Non-tuberculosis Mycobacteria (NTM) Lung Disease
Description: Number of patients with non-tuberculosis mycobacteria (NTM) lung disease is reported. NTM lung disease was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for NTM recorded as any diagnosis during the following period after the index date.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
Participants | 27 | 14
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.1158, Regression, Cox; Hazard Ratio (HR) = 0.590, 95% CI 2-sided [0.305 to 1.139]

49. Secondary Outcome: Time to Non-tuberculosis Mycobacteria (NTM) Lung Disease From the Index Date
Description: Median and Inter-Quartile Range of Time to non-tuberculosis mycobacteria (NTM) lung disease from the index date were estimated using the Kaplan-Meier curve.
  NTM lung disease was defined as ≥1 inpatient claims or outpatient claims 1) with ICD-10 codes for NTM recorded as any diagnosis during the following period after the index date.
  Date of NTM was defined as the admission date of inpatient claim or the starting date of outpatient claim with the above 1 condition to define NTM event.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | LAMA | ICS/LABA
Number analyzed (Participants) | 2444 | 2444
days | 129 [49 to 815] | 360.5 [99 to 612]
Statistical Analysis 1: Comparison: LAMA vs ICS/LABA; Test type: Other; p = 0.11, Log Rank

ADVERSE EVENTS:
Time Frame: All-Cause-mortality: From the index date (i.e. between 01 January 2005 and 30 April 2015) up to the earliest of discontinuation of the index drug (i.e. LAMA or ICS/LABA), death, or 30 April 2016 (i.e. cut-off date for data retrieving), up to 136 months.
Description: This is a non-interventional study using national health insurance claims data from the National Health Insurance Service (NHIS). No adverse events were collected on an individual case level.
  Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
  All-Cause Mortality is an outcome of this study and thus additionally reported below.
Groups:
- LAMA: Chronic obstructive pulmonary disease (COPD) patients who were prescribed long-acting muscarinic antagonists (LAMA) monotherapy between 01 January 2005 and 30 April 2015.
  Participants were matched 1:1 ('LAMA' : 'ICS/LABAs') using propensity scores estimated as by multiple logistic regression analysis based on age, sex, socioeconomics status, Charlson Comorbidity Index, asthma and history of chronic obstructive pulmonary disease (COPD) exacerbation.
- ICS/LABA: Chronic obstructive pulmonary disease (COPD) patients who were prescribed a fixed-dose combination (FDC) of inhaled corticosteroid (ICS)/long-acting beta agonists (LABA) between 01 January 2005 and 30 April 2015.
  Participants were matched 1:1 ('LAMA' : 'ICS/LABAs') using propensity scores estimated as by multiple logistic regression analysis based on age, sex, socioeconomics status, Charlson Comorbidity Index, asthma and history of chronic obstructive pulmonary disease (COPD) exacerbation.
Arm/Group | LAMA | ICS/LABA
All-Cause Mortality (participants affected / at risk) | 51/2444 | 46/2444
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT04172701/Prot_SAP_000.pdf